CLINICAL TRIAL: NCT05295680
Title: A Study of Oral Hymecromone to Treat Adolescents and Adults With Primary Sclerosing Cholangitis(HAAPS Study).
Brief Title: Oral Hymecromone to Treat Adolescents and Adults With Primary Sclerosing Cholangitis.
Acronym: HAAPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aparna Goel (Other)
Responsible Party: Sponsor-Investigator, Aparna Goel, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64030
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-11

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Hymecromone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hymecromone (Experimental): Participants will receive Hymecromone for six months + Standard Of Care (SOC), and will be followed for an additional nine months.
  Interventions: Drug: Hymecromone
- Standard Of Care (SOC) (No Intervention): Participants will receive Standard Of Care (SOC), and will be followed for 15 months.

INTERVENTIONS:
Drug: Hymecromone — Hymecromone 400 mg 3 times daily by mouth.
  Other Names: Isochol
  Arms: Hymecromone

SUMMARY:
Primary objective: To evaluate the efficacy of hymecromone plus standard of care compared with standard of care alone in the treatment of adolescents and adults with primary sclerosing cholangitis (PSC).

Secondary objectives: To evaluate the change in Alkaline Phosphatase (ALP) from baseline to 6 months post-treatment following treatment with hymecromone plus standard of care compared with standard of care.

To evaluate changes in biomarkers of PSC disease during hymecromone treatment, namely: (a) fibrotic effect (FibroScan); (b) inflammatory biomarkers (serum Hyaluronan (HA)); and, (c) T-cell count.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary sclerosing cholangitis confirmed by liver biopsy and/or imaging study
* If history of endoscopically confirmed inflammatory bowel disease, currently stable based on Mayo Score / Disease Activity Index (DAI) for Ulcerative Colitis Score ≤ 1, normal inflammatory markers (ESR, CRP and fecal calprotectin) and stable non-excluded medical therapy for at least 6 months

Exclusion Criteria:

* Currently receiving biologic therapies
* Known allergy to hymecromone
* Cholangiocarcinoma
* Pregnancy
* Serious liver disease

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum gamma-glutamyltransferase (GGT) levels | Baseline to Month 6

SECONDARY OUTCOMES:
Change in serum Alkaline Phosphatase (ALP) levels | Baseline to Month 6
Change in serum hyaluronan levels | Baseline to Month 6
Change in T-cell count | Baseline to Month 6
Change in fibrotic effect based on FibroScan | Baseline to Month 6
  Fibrotic effect is the amount of liver with fatty change
Change in biliary tree anatomy (e.g. strictures) based on FibroScan | Baseline to Month 6
Change in serum inflammatory cytokine profile | Baseline to Month 6
  This outcome measure will assess pro-inflammatory cytokines previously associated with biliary inflammation and other autoimmune diseases including IFNg, IL-6, and TNF.
Change in lymphocyte immunophenotype | Baseline to Month 6
  Single cell analysis technique will be used to assess the lymphocytes (B- and T-cells) present in serum samples, including FoxP3+ regulatory T-cells, a tolerogenic lymphocyte subset with important roles in immune tolerance.
Plasma drug levels of 4-MU | Single blood draw at baseline, week 2, and months 1, 3, and 6 study visits
Plasma drug levels of 4-MUG | Single blood draw at baseline, week 2, and months 1, 3, and 6 study visits
Plasma drug levels of 4-MUS | Single blood draw at baseline, week 2, and months 1, 3, and 6 study visits

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Goel, MD, Principal Investigator — Stanford University; Leina Alrabadi, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Clinic, Redwood City, California
  - Stanford Clinic, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salman L, Martinez L, Faddoul G, Manning C, Ali K, Salman M, Vazquez-Padron R. Hyaluronan Inhibition as a Therapeutic Target for Diabetic Kidney Disease: What Is Next? Kidney360. 2023 Jun 1;4(6):e851-e860. doi: 10.34067/KID.0000000000000126. Epub 2023 Apr 14. PMID 37055910